CLINICAL TRIAL: NCT00913328
Title: Effect of Add-on Montelukast to Inhaled Corticosteroids in Excessive Airway Narrowing in Adults With Asthma
Brief Title: Effect of Add-on Montelukast to Inhaled Corticosteroids on Airway Responsiveness
Acronym: SINGDEN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Ass. prof. of Medicine Charlotte Suppli Ulrik, Department of Heart and Lung Diseases, Hvidovre Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SINGDEN-04-2002
Record Dates: First submitted 2009-06-03; First posted 2009-06-04 (Estimated); Last update posted 2009-06-04 (Estimated); Status verified 2009-06

CONDITIONS: Asthma
Keywords: Asthma; Airway responsiveness; Dose-response plateau; Montelukast; Add-on to inhaled corticosteroids
MeSH Terms: conditions — Asthma | interventions — montelukast

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Montelukast (Active Comparator): Oral montelukast 10 mg once daily for 12 weeks
  Interventions: Drug: Montelukast (Singulair)
- Placebo (Placebo Comparator): Oral placebo once daily for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Montelukast (Singulair) — 10 mg tablet once daily
  Other Names: Singulair
  Arms: Montelukast
Drug: Placebo — Oral placebo once daily
  Arms: Placebo

SUMMARY:
Leukotriene receptor antagonists appear to posses additive anti-inflammatory effects to the effect of inhaled corticosteroids.

Hypothesis: Treatment with oral montelukast will lower the dose-response plateau to inhaled methacholine in patients with mild to moderate persistent asthma treated with a stable dose of inhaled corticosteroids.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoking adults with mild to moderate persistent asthma:

  * FEV1 > 70 % pred
  * PD20 methacholine < 3.9 mmol
  * treated for at least 3 months with a stable dose of inhaled corticosteroids
* Documented dose-response plateau to inhaled methacholine on two occasions
* Males and non-pregnant females

Exclusion Criteria:

* Asthma medication other than inhaled corticosteroids and inhaled b2-agonists
* Viral respiratory tract infections within the 3 weeks prior to enrollment

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2002-08; Primary Completion 2006-05 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in maximal FEV1 decline at the dose-response plateau | After 12 weeks of treatment

SECONDARY OUTCOMES:
Changes from baseline in PD20 methacholine | After 12 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Zuzana Diamant, MD, PhD, Principal Investigator — Erasmus Medical Center; Charlotte S Ulrik, MD, DMSc, Principal Investigator — Dept. of Heart and Lung Diseases, Hvidovre Hospital, Denmark